CLINICAL TRIAL: NCT02182258
Title: Safety and Tolerability of Single Rising Doses of 1 mg, 3 mg, 10 mg and 20 mg of BIBF 1120 as Intravenous Infusion (Single-blind, Placebocontrolled at Each Dose Group) and Absolute Bioavailability of 100 mg BIBF 1120 as Soft Gelatine Capsule (Intra-individual Comparison)
Brief Title: Safety and Tolerability Study of BIBF 1120 as Intravenous Infusion and Absolute Bioavailability of BIBF 1120 as Soft Gelatine Capsule in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1199.75
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo ampoule
- BIBF 1120 intravenous (Active Comparator)
  Interventions: Drug: BIBF 1120 intravenous solution
- BIBF 1120 capsule (Experimental)
  Interventions: Drug: BIBF 1120 soft gelatine capsule

INTERVENTIONS:
Drug: BIBF 1120 soft gelatine capsule
  Arms: BIBF 1120 capsule
Drug: BIBF 1120 intravenous solution
  Arms: BIBF 1120 intravenous
Drug: Placebo ampoule
  Arms: Placebo

SUMMARY:
The primary objective of this trial was to assess the safety and tolerability of BIBF 1120 administered as intravenous (iv) infusions of 1, 3, 10, and 20 mg, and to assess the absolute bioavailability of orally administered 100 mg BIBF 1120 as soft gelatine capsules. A secondary objective was the exploration of the pharmacokinetic (PK) of BIBF 1120 after single iv dosing, including dose proportionality.

ELIGIBILITY:
Inclusion Criteria:

Healthy males according to the following criteria:

1. Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate), 12-lead ECG, and clinical laboratory tests
2. Age ≥18 years and ≤50 years
3. Body mass index (BMI) ≥18.5 and ≤29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

Exclusion Criteria:

1. Any finding from medical examination (including blood pressure, pulse rate, ECG) deviating from normal and of clinical relevance
2. History of or current gastrointestinal, hepatic (including Gilbert's syndrome and history of bilirubin increases) renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
3. History of relevant orthostatic hypotension, fainting spells, and blackouts
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy or its excipients) which is deemed relevant to the trial as judged by the investigator
7. History of any bleeding disorder including prolonged or habitual bleeding, other haematologic disease or cerebral bleeding (e.g. after a car accident) or commotio cerebri
8. Intake of drugs with a long half-life (>24 h) within 1 month prior to administration or during the trial
9. Use of any drugs which might influence the results of the trial within 14 days prior to administration or during the trial
10. Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
11. Smoker (>10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
12. Alcohol abuse (>30 g/day)
13. Drug abuse
14. Blood donation (>150 mL within 4 weeks prior to administration or during the trial)
15. Excessive physical activities within 5 days prior to administration or during the trial
16. Any laboratory value outside the reference range that is of clinical relevance
17. Male subjects refusing to minimise the risk of female partners becoming pregnant from the first dosing day until 3 months after completion of the study. Acceptable methods of contraception for male volunteers include vasectomy no less than 3 months prior to administration, barrier contraception, or a medically accepted contraceptive method. Acceptable methods of contraception for female partners of male volunteers include intra-uterine device, tubal ligation, hormonal contraceptive for at least 2 months and diaphragm with spermicide.
18. Homozygous genotype status for UGT1A1*28, *60 (Gilbert polymorphisms)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 48 hours after drug administration
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) | Up to 48 hours after drug administration

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 48 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | Up to 48 hours after drug administration
%AUCtz-∞ (calculated from AUC0-∞ and AUC0-tz ) | Up to 48 hours after drug administration
Terminal rate constant in plasma (λz) | Up to 48 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | Up to 48 hours after drug administration
Mean residence time of the analyte in the body after oral administration (MRTpo) | Up to 48 hours after drug administration
Mean residence time of the analyte in the body after iv administration (MRT) | Up to 48 hours after drug administration
Apparent clearance of the analyte in plasma after extravascular administration (CL/F) | Up to 48 hours after drug administration
Apparent clearance of the analyte in plasma after intravenous administration (CL) | Up to 48 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | Up to 48 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an intravenous dose (Vz) | Up to 48 hours after drug administration
Apparent volume of distribution at steady-state following an intravenous dose (Vss) | Up to 48 hours after drug administration
Amount of analyte that is eliminated in urine within the time interval t1 to t2 (Aet1-t2) | Up to 48 hours after drug administration
Fraction of analyte excreted in urine within the time interval t1 to t2, in percentage of dose (fet1-t2) | Up to 48 hours after drug administration
Renal clearance of analyte within the time interval t1 to t2 (CLR,t1-t2) | Up to 48 hours after drug administration
Change from baseline in physical examination | Baseline, day 46
Change from baseline in vital signs (BP, PR) | Baseline, day 46
Change from baseline in 12-lead ECG (electrocardiogram) | Baseline, day 46
Change from baseline in clinical laboratory test (hematology, clinical chemistry and urinalysis) | Baseline, day 46
Number of Participants with Serious and Non-Serious Adverse Events | Up to day 46
Assessment of tolerability by investigator on a four point scale (good, satisfactory, not satisfactory, bad) | Up to day Day 46